CLINICAL TRIAL: NCT02287415
Title: The Effect of BIA 2-093 on the Steady-state Pharmacodynamic and Pharmacokinetic Profiles of Warfarin in Healthy Volunteers
Brief Title: The Effect of BIA 2-093 on the Steady-state Pharmacodynamic and Pharmacokinetic Profiles of Warfarin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-108
Record Dates: First submitted 2014-11-06; First posted 2014-11-10 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 (Experimental): Phase A: Warfarin Phase B: Warfarin + BIA 2-093 (ESL) Phase C: Warfarin
  Interventions: Drug: BIA 2-093; Drug: Warfarin

INTERVENTIONS:
Drug: BIA 2-093
  Other Names: ESL, Eslicarbazepine acetate
Drug: Warfarin
  Other Names: Uniwarfin

SUMMARY:
Multiple-dose, open-label, single-period study consisting of three consecutive phases

DETAILED DESCRIPTION:
Multiple-dose, open-label, single-period study consisting of three consecutive phases: Phase A - run-in warfarin dose-finding phase Phase B - warfarin pharmacokinetics (PK) and international normalised ratio (INR) profiling Phase C - warfarin alone at their individualised doses

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 18 and 45 years, inclusive
* Subjects of body mass index (BMI) between 19 and 28 kg/m2, inclusive
* Subjects who were healthy as determined by pre-study medical history, physical examination, neurological examination, and 12-lead ECG
* Subjects who had clinical laboratory tests clinically acceptable
* Subjects who were negative for HBs Ag, anti-HCV Ab and anti-HIV-1 and HIV-2 Ab tests at screening
* Subjects who were negative for alcohol and drugs of abuse at screening
* Subjects who were non-smokers or who smoked less than 10 cigarettes or equivalent per day
* Subjects who were able and willing to give written informed consent
* In case of female volunteers, subjects who were not of childbearing potential by reason of surgery or, if of childbearing potential, used one of the following methods of contraception: double-barrier or intrauterine device
* In case of female volunteers, subjects who had a negative pregnancy test at screening

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria
* Subjects who had a clinically relevant history or presence of respiratory gastrointestinal, renal, hepatic, haematological, lymphatic, neurological cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological dermatological, endocrine, connective tissue diseases or disorders
* Subjects who had a current haemostatic disorder or a personal or family history of any such disorder
* Subjects who had a personal or family history of bleeding complications after surgery or tooth extraction, nose or gingival bleeding, or haemorrhagic diathesis.
* Subjects with a profession or activities implying a special risk of trauma
* Subjects with any abnormality in the coagulation status (aPTT or prothrombin INR)
* Subjects who had a clinically relevant surgical history
* Subjects who had a clinically relevant family history
* Subjects who had a history of relevant atopy
* Subjects who had a history of relevant drug hypersensitivity
* Subjects who had a history of alcoholism or drug abuse
* Subjects who consumed more than 14 units of alcohol a week
* Subjects who had a significant infection or known inflammatory process on screening and/or admission
* Subjects who had acute gastrointestinal symptoms at the time of screening and/or admission (e.g., nausea, vomiting, diarrhoea, heartburn)
* Subjects who had used prescription drugs within 2 weeks prior admission on Phase A
* Subjects who had used any investigational drug and/or participated in any clinical trial within 2 months prior admission to Phase A
* Subjects who had previously received BIA 2-093
* Subjects who had donated and/or received any blood or blood products within the previous 2 months prior admission to Phase A
* Subjects who were vegetarians, vegans and/or had medical dietary restrictions
* Subjects who could not communicate reliably with the investigator

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2002-05; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Phase A: Warfarin Phase B: Warfarin + BIA 2-093 (ESL) Phase C: Warfarin
  BIA 2-093
  Warfarin
Period: Overall Study
Arm/Group | Group 1
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Group 1
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Steady-state Plasma Concentration
Time Frame: PHASE A: first 3 days; PHASE B: Days 1, 2, 4, 6, 7 and 8: pre-dose. PHASE C: Days 1, 3, 5 and 7: pre-dose; Day 8: 24 h post last-warfarin dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Group 1
Number analyzed (Participants) | 13
ng/mL | 31652 (11150)

2. Secondary Outcome: Tmax - Time of Occurrence of Cmax
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1
Number analyzed (Participants) | 13
hours | 6 [1 to 12]

3. Secondary Outcome: AUCτ - Steady-state Area Under the Plasma Concentration-time Profile Over 24 h, the Dosing Interval
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Group 1
Number analyzed (Participants) | 13
ng.h/mL | 411834 (113305)

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 9/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=13)
Lymphadenopathy inguinal (Blood and lymphatic system disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Lumbago (Musculoskeletal and connective tissue disorders) | 1
Pain in elbow (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Tension headache (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Vasovagal reaction (Nervous system disorders) | 1
Lipothymia (Nervous system disorders) | 1
Irritability (Psychiatric disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Adhesive tape allergy (Skin and subcutaneous tissue disorders) | 1
Hot flashes (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes